CLINICAL TRIAL: NCT01507012
Title: A Double Blind, Placebo Controlled Study Measuring The Effect Of Berry Polyphenols On Mood And Cognition In Healthy Adults
Brief Title: The Effect Of Berry Polyphenols On Human Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: The New Zealand Institute of Plant and Food Research Ltd. (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 28AI1
Record Dates: First submitted 2011-09-20; First posted 2012-01-10 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Berry phenolics; mood; cognition; adults

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Powdered berryfruit extract (Experimental): Powdered berry extract containing 500mg of polyphenols
  Interventions: Dietary Supplement: Berry Polyphenols
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Berryfruit juice (Experimental): Berryfruit juice containing 500mg polyphenols
  Interventions: Dietary Supplement: Berry Polyphenols

INTERVENTIONS:
Dietary Supplement: Berry Polyphenols
  Arms: Berryfruit juice; Powdered berryfruit extract
Dietary Supplement: Placebo — Placebo control containing sugar and artificial flavouring.
  Arms: Placebo

SUMMARY:
Polyphenols, compounds found at high levels in berry fruit, have been shown to have health promoting benefits through various mechanisms both in vivo and in vitro. These benefits include antioxidant activity, anti-inflammatory properties, and monoamine oxidase (MAO) inhibition. This study aims to expand on the extremely promising animal data in the literature, and our own pilot study results, to investigate whether drinks containing berry fruit can improve cognitive performance and mood in healthy human participants.

Our central hypothesis is that fruit extracts can reduce the breakdown of neurotransmitters such as dopamine and serotonin. This reduction in breakdown could therefore increase the levels of these neurotransmitters and convey some benefits in regards to mood and cognitive function. The investigators will assess the pharmacokinetic activity of berry fruit extracts on MAO activity to test this hypothesis.

A second hypothesis is that berryfruit polyphenols may alter circulating levels of glucose that may in turn affect cognitive performance and mood.

A prior study carried out by Plant & Food Research through collaboration with the University of Northumbria, UK, found promising results after acutely supplementing participants with a berry fruit based drink. This study aims to use the results from the previous study to assess in depth the effect of berry fruit drinks on human behaviour.

DETAILED DESCRIPTION:
This project will investigate the acute effects on human cognitive behaviour and mood of a single consumption of 2 berryfruit drinks (with balanced polyphenol content) versus a placebo. Drinks are matched for taste, sugar content and appearance. Drinks contain natural berry fruit grown and juiced or extracted in New Zealand under food-safe conditions.

The study will follow a double-blind, counterbalanced, placebo controlled, repeated measures design with 36 healthy participants aged between 18 and 30 completing 3 study day sessions as well as one training/screening visit (four visits in total). On one occasion participants will receive a placebo, on another berryfruit drink 1, and on another berryfruit drink 2. Study days will be spaced one week apart to accommodate a wash out period. Both berryfruit drinks will be made to include 500mg of polyphenols/60kg of body weight. Sucralose (artificial sweetener) will be added to make the drinks palatable. Participants will be screened for any intolerance or allergies to the drinks during the training/screening session.

Psychometric tasks and mood scales will be measured using the Computerised Mental Performance Assessment System (COMPASS), a purpose designed software application for the flexible delivery of randomly generated parallel versions of standard and novel cognitive assessment tasks that has previously been shown to be sensitive to nutritional interventions and was used in the prior study conducted at Northumbria University. The cognitive assessment battery will include: Bond-Lader mood scales, visual analogue mood scales, 7 repetitions of Digital Vigilance, Stroop, Rapid Visual Information Processing and Mental Fatigue Visual Analogue scales. This is followed by a logical reasoning task and a final set of the Bond-Lader mood scales.

Baseline cognitive testing will involve one repetition of the cognitive assessment battery (Bond-Lader mood scales, Visual Analogue scales, Digital Vigilance, Stroop and RVIP followed by a second set of Visual Analogue scales).

On all 3 testing days participants will arrive at the lab in the morning (8:30 am), after an overnight fast, and firstly give a 10 mL venous blood sample taken by a trained phlebotomist. Participants will then have their blood glucose measured via a finger prick and heart rate/blood pressure (autonomic measures) measured using an automated digital blood pressure monitor. Participants will then complete one repetition of the COMPASS computerised cognitive assessment battery (baseline). Participants will then be orally supplemented with treatment in the form of a single serve juice drink.

After a 60 minute absorption period, autonomic measurements and a second blood glucose reading will be taken. Participants will then complete the COMPASS assessment. After completion of the assessment, a third set of autonomic measurements will be immediately taken along with a third blood glucose reading and a second 10 mL venous blood sample.

ELIGIBILITY:
Inclusion Criteria:

* MMale/female,
* Healthy Age 18-35 years old
* Non smoker
* Proficient in English
* Not taking any herbal or prescription medications
* Not pregnant or seeking to become pregnant, BMI < 30kg/m2

Exclusion Criteria:

* Tobacco user,
* pregnant or seeking to become pregnant,
* currently taking recreational over the counter/prescription medication (excluding the contraceptive pill) and/or dietary/herbal supplements.
* Food allergies or sensitivities that are relevant to the study,
* learning difficulties,
* ADHD,
* dyslexia,
* migraines or
* any gastric problems

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Attention and vigilance | baseline, 1 hour post dose then incrementally every 10 minutes for 70 minutes.
  Attention and vigilance will be measured at baseline ad then 1 hour post supplementation of the study treatment. at baseline the digit vigilance task, stroop task and RVIP task will be completed. One hour post supplementation of the study treatment, 7 sets of digit vigilance, stroop and RVIP will be completed. The outcome measures will be treated as change from baseline scores.
Change from baseline blood platelet monoamine oxidase-B activity | Baseline and 150 minutes post dose
Change from baseline visual analogue scale fatigue | baseline, 1 hour post dose then incrementally every 10 minutes for 70 minutes.
Change from baseline blood glucose mmol/L | Baseline, 60 minutes post dose and 150 minutes post dose
Change from baseline blood plasma anthocyanin levels | Baseline and 150 minutes post supplementation
Change from baseline visual analogue scale difficulty | baseline, 1 hour post dose then incrementally every 10 minutes for 70 minutes.
Change from baseline Bond Lader mood scales | Baseline, 60 minutes and 1 hour 50 minutes post dose
Change from baseline diastolic blood pressure | Baseline, 60 minutes and 150 minutes
Change from baseline systolic blood pressure | Baseline, 60 minutes and 150 minutes post supplementation
Change from baseline logical reasoning | Baseline and 150 minutes post supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Anthony W Watson, Principal Investigator — Northumbria University
Locations (1):
- The New Zealand Institute for Plant & Food Research Ltd, Auckland, New Zealand